CLINICAL TRIAL: NCT04197310
Title: Phase II Trial of Cabozantinib in Combination With Nivolumab for Advanced Carcinoid Tumors
Brief Title: Cabozantinib and Nivolumab for Carcinoid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry); Exelixis (Industry)
Responsible Party: Principal Investigator, Kimberly Perez, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-403
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Results first posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Carcinoid Tumor; Carcinoid Tumor of GI System; Neuroendocrine Tumors
Keywords: Carcinoid Tumor; Carcinoid Tumor of GI System; Neuroendocrine Tumors
MeSH Terms: conditions — Carcinoid Tumor; Neuroendocrine Tumors | interventions — Nivolumab; cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab and Cabozantinib (Experimental): The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.
  * Cabozantinib will be administered at a dose of 40mg orally, once daily
  * Nivolumab will be given at a dose of 240mg every 14 days, intravenously
  Retreat Phase (Optional)
  * Participants may elect to stop nivolumab and cabozantinib with confirmed CR after at least 24 weeks of treatment.
  * Participants who elect to stop and then the condition progresses after stopping study treatment may be eligible to resume nivolumab and cabozantinib therapy.
  * This resumption will be termed as a retreatment second course phase and is available only while the study remains open and the subject meets specified criteria.
  Interventions: Drug: Nivolumab; Drug: Cabozantinib

INTERVENTIONS:
Drug: Nivolumab — 240mg, intravenously, Day 1 and 15 of a 28 day cycle
  Other Names: Opdivo
Drug: Cabozantinib — 40mg, orally, Daily for a 28 day cycle
  Other Names: Cometriq; Cabometyx

SUMMARY:
This research study, is studying the combination of cabozantinib and nivolumab in treating advanced carcinoid tumors.

- Carcinoid tumor is another term used to refer to neuroendocrine tumors that arise in organs such as the gastrointestinal tract, lungs, or thymus.

DETAILED DESCRIPTION:
This is open-label, single-arm, phase II research study, studying the combination of cabozantinib and nivolumab in treating advanced carcinoid tumors. Carcinoid tumor is another term used to refer to neuroendocrine tumors that arise in organs such as the gastrointestinal tract, lungs, or thymus.

* The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.
* Cabozantinib will be administered orally, once daily
* Nivolumab will be administered intravenously, every two weeks
* The target enrollment for this study is 35 participants.
* The U.S. Food and Drug Administration (FDA) has not approved cabozantinib or nivolumab for treating carcinoid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally unresectable or metastatic well-differentiated neuroendocrine tumor of non-pancreatic (ie, carcinoid) origin
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan, MRI, or calipers by clinical exam. See Section 11 for the evaluation of measurable disease.
* Patients must have evidence of radiographic disease progression within the past 12 months.
* Patients who have received at least one line of therapy, which can include somatostatin analog therapy. Participants should be adequately recovered from acute toxicities of prior treatment.

  * Prior somatostatin analog therapy is allowed. Continuation of somatostatin analog therapy is allowed provided that the dose has been stable for 2 months.
  * Prior chemotherapy: Participants must have been off treatment with cytotoxic chemotherapy for at least 14 days prior to registration.
  * Prior biologic therapy: Patients must have discontinued all biologic therapy at least 28 days prior to registration. Duration may be shorted to 14 days for agents with short half-lives.
  * Prior radiolabeled somatostatin analog therapy: Participants must have completed radiolabeled somatostatin analog therapy at least 6 weeks prior to registration.
  * Prior hepatic artery embolization or ablative therapies is allowed if measurable disease remains outside the treated area or there is documented disease progression in a treated site. Prior liver-directed or ablative treatment must be completed at least 28 days prior to registration.
  * Prior radiation therapy: Radiation therapy must be completed per the following timelines

    * i) Radiotherapy to the thoracic cavity or abdomen within 4 weeks prior to registration.
    * ii) Radiotherapy to bone lesions within 2 weeks prior to registration.
    * iii) Radiotherapy to any other site within 4 weeks prior to registration.
    * NOTE: In all cases, there must be complete recovery and no ongoing complications from prior radiotherapy.
* Age ≥ 18 years.
* ECOG performance status ≤1 (Karnofsky ≥60%, see Appendix A)
* Participants must have normal organ and marrow function as defined below:

  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * total bilirubin ≤1.5 × institutional upper limit of normal (ULN) (or 2.0 x ULN in patients with documented Gilbert's Syndrome)
  * AST (SGOT)/ALT (SGPT) ≤2.5 × ULN or ≤ 3 × ULN for participants with documented liver metastases
  * creatinine <1.5 × ULN Or creatinine clearance ≥40 mL/min (using Cockcroft-Gault formula) for participants with creatinine levels above institutional normal
  * Urine protein/creatinine ratio (UPCR) ≤ 1
  * PT/INR or partial thromboplastin time (PTT) test < 1.3 the laboratory ULN within 7 days before the first dose of study treatment.
* Negative urine pregnancy test for women of childbearing potential.
* Participant must be able to swallow pills.
* The participant is capable of understanding and complying with the protocol and has signed the informed consent document.

Exclusion Criteria:

* Major surgery (eg, GI surgery, removal or biopsy of brain metastasis) within 8 weeks before first dose of study treatment. Complete wound healing from major surgery must have occurred 1 month before first dose and from minor surgery (eg, simple excision, tooth extraction) at least 10 days before first dose. Subjects with clinically relevant ongoing complications from prior surgery are not eligible.
* Participants who are receiving any other investigational agents.
* Participants who have received a prior cabozantinib.
* Participants who have received prior therapy with an anti-PD-1, anti-PD-L1, anti- PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including nivolumab, pembrolizumab, ipilimumab, and any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* The participant has tumor in contact with, invading, or encasing major blood vessels or radiographic evidence of significant cavitary pulmonary lesions.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cabozantinib or nivolumab.
* Participants receiving any strong inhibitors or inducers of CYP3A4 within 14 days prior to registration are ineligible. Chronic treatment with strong inhibitors or inducers of CYP3A4 is not allowed.
* Cardiovascular disorders including:

  * Congestive heart failure (CHF): New York Heart Association (NYHA) Class III (moderate) or Class IV (severe) at the time of screening;
  * Concurrent uncontrolled hypertension defined as sustained blood pressure (BP) > 150 mm Hg systolic or > 100 mm Hg diastolic despite optimal antihypertensive treatment within 7 days of the first dose of study treatment;
  * Any history of congenital long QT syndrome;
  * QTcF interval >500 msec
  * Any of the following within 6 months before the first dose of study treatment:

    * unstable angina pectoris;
    * clinically-significant cardiac arrhythmias;
    * stroke (including transient ischemic attack (TIA), or other ischemic event);
    * myocardial infarction;
* GI disorders particularly those associated with a high risk of perforation or fistula formation including:

  * Tumors invading the GI tract, active peptic ulcer disease, active inflammatory bowel disease (eg, Crohn's disease), active diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis or acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction
  * Abdominal fistula, GI perforation, bowel obstruction, intra-abdominal abscess within 6 months before screening
* Thromboembolic events within 6 months of registration.

  * Note: Low dose aspirin ≤ 81 mg/day is allowed. Anticoagulation with therapeutic doses of LMWH is allowed in patients who are on a stable dose of LMWH for at least 6 weeks prior to registration. Treatment with warfarin is not allowed.
* The subject has experienced any significant bleeding episodes, including:

  * Clinically significant gastrointestinal bleeding within 6 months before the first dose of study treatment
  * Clinically significant hemoptysis (> 0.5 teaspoon) within 3 months of the first dose of study treatment
  * Any other signs indicative of pulmonary hemorrhage within 3 months before the start of study treatment
  * Individuals with a history of different malignancy are ineligible except for the following circumstances: Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years or are deemed by the investigator to be at low risk for recurrence of that malignancy.
* Participant has an active infection requiring IV antibiotics
* Any active, known, or suspected autoimmune disease. Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (e.g. celiac disease) are permitted to enroll.
* Patient has a medical condition that requires chronic systemic steroid therapy or on any other form of immunosuppressive medication. Adrenal replacement steroid disease are permitted in the absence of autoimmune disease.
* The participant is known to be positive for the human immunodeficiency virus (HIV), HepBsAg, or HCV RNA. HIV-positive participants with non-detectable viral loads on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with cabozantinib and nivolumab.
* The participant has received a live vaccine within 28 days prior to the first dose of trial treatment and while participating in the trial. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, BCG, and typhoid vaccine. The use of the inactivated seasonal influenza vaccine (Fluzone®) is allowed.
* Pregnant or lactating females are excluded from this study because cabozantinib and nivolumab are agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with cabozantinib and nivolumab, breastfeeding should be discontinued if the mother is treated with cabozantinib and nivolumab. These potential risks may also apply to other agents used in this study.
* Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (eg, barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and following treatment. Women of childbearing potential receiving nivolumab will be instructed to adhere to contraception for a period of 5 months after the last dose of nivolumab. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose of nivolumab. Contraception must be used for 4 months after last dose of cabozantinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-12-26 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Perez, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Boston Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivolumab + Cabozantinib: The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.
  * Cabozantinib will be administered at a dose of 40mg, orally, once daily for a 28 day cycle
  * Nivolumab will be given at a dose of 240mg, intravenously, Day 1 and 15 of a 28 day cycle
Period: Overall Study
Arm/Group | Nivolumab + Cabozantinib
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were collected for all participants enrolled on the study (19)
Arm/Group | Nivolumab + Cabozantinib
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined by RECIST 1.1 criteria, the percentage of subjects with a confirmed complete response or partial response at any time during treatment. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the diameters of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 46 months
Measure: Number; unit: percentage of participants
Arm/Group | Nivolumab + Cabozantinib
Number analyzed (Participants) | 19
percentage of participants | 0

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-Free Survival (PFS) is defined as the time from randomization (or registration) to the earlier of progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesion and/or unequivocal progression of existing non-target lesions are also considered progression. Unequivocal progression should not normally trump target lesion status and must be representative of overall disease status change, not a single lesion increase.
Time Frame: Time from randomization (or registration) to the earlier of progression or death due to any cause. The median survival follow-up time was 5.6 months (range 1.4 - 31.0 months).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab + Cabozantinib
Number analyzed (Participants) | 19
months | 5.6 [3.5 to 9.9]

3. Secondary Outcome: Overall Response Rate (ORR) Per Immune-related Response Criteria
Description: ORR will be determined according to immune-related response criteria (irRC). irComplete Response (irCR): Complete disappearance of all target lesions. irPartial Response (irPR): Decrease, relative to baseline, or 50% or greater in the sum of the products of the two largest perpendicular diameters of all target and all new measurable target lesions. irStable Disease (irSD): Does not meet criteria for irRC or irPR, in the absence of progressive disease. irProgressive Disease (irPD): At least 25% increase Percentage Change in Tumor Burden when compared to SPD at nadir.
Time Frame: 46 months
Population: A total of 17 participants were analyzed for ORR using irRC, with data from 2 participants unavailable for analysis based on this criterion.
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Cabozantinib
Number analyzed (Participants) | 17
Participants | 0

4. Secondary Outcome: Overall Survival (OS)
Description: Kaplan and Meier to assess Overall survival (OS).
Time Frame: Overall Survival (OS) is defined as the time from randomization (or registration) to death due to any cause, or censored at date last known alive. OS was calculated for a median of 6.9 months, ranging from 2.8 - 31.0 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab + Cabozantinib
Number analyzed (Participants) | 19
months | 16.0 [6.5 to NA] — The upper limit of the 95% confidence interval was not detected due to an insufficient number of participants with events.

5. Secondary Outcome: Number of Participants With Treatment Related Adverse Events
Description: Safety was assessed by analysis of adverse event (AE) and toxicity data. AE and toxicity data are defined according to NCI CTCAE version 5.0. Adverse Events were reviewed between the initial dose of study treatment and 100 days of the last dose of treatment. All adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv5 as reported on case report forms will be counted. Rate is the proportion of treated participants experiencing at least one treatment-related AE of any type during the time of observation.
Time Frame: AEs were reviewed between the initial dose of study treatment and 100 days of the last dose of treatment. AEs were assessed for a median of 8.8 months, ranging from 4.7 - 33.7 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Cabozantinib
Number analyzed (Participants) | 19
Participants | 19

6. Secondary Outcome: Duration of Response
Description: To evaluate duration of response of participants receiving Nivolumab and Cabozatinib. Duration of response was evaluated from date of registration to date of death or last known date alive.
Time Frame: The median survival follow-up time was 5.6 months (range 1.4 - 31.0 months).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab + Cabozantinib
Number analyzed (Participants) | 19
months | NA [NA to NA] — Duration of response was not observed due to a lack of participants with events.

ADVERSE EVENTS:
Time Frame: Adverse events were recorded between the first patient treated (March 2020) and 100 days out from the last patient ending treatment (December 2023). Participants were assessed for AEs for a median of 8.8 months (range 4.7 - 33.7 months)
Description: Adverse events were reviewed and reported after the initial dose of study treatment, during treatment, or within 100 days of the last dose of treatment.
Arm/Group | Nivolumab + Cabozantinib
All-Cause Mortality (participants affected / at risk) | 8/19
Serious Adverse Events (participants affected / at risk) | 9/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Cabozantinib (N=19)
Abdominal pain (Gastrointestinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 3
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 3
Colitis (Gastrointestinal disorders) | 1
Confusion (Psychiatric disorders) | 3
Constipation (Gastrointestinal disorders) | 1
Creatinine increased (Investigations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Renal calculi (Renal and urinary disorders) | 1
Seizure (Nervous system disorders) | 1
Sepsis (Infections and infestations) | 2
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Cabozantinib (N=19)
Abdominal pain (Gastrointestinal disorders) | 9
Agitation (Psychiatric disorders) | 1
Alanine aminotransferase increased (Investigations) | 15
Alkaline phosphatase increased (Investigations) | 12
Anemia (Blood and lymphatic system disorders) | 11
Anorexia (Metabolism and nutrition disorders) | 9
Anxiety (Psychiatric disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Ascites (Gastrointestinal disorders) | 1
Aspartate aminotransferase increased (Investigations) | 14
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bloating (Gastrointestinal disorders) | 2
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1
Blood bicarbonate decreased (Investigations) | 1
Blood bilirubin increased (Investigations) | 5
Blood lactate dehydrogenase increased (Investigations) | 1
Blurred vision (Eye disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 3
Bruising (Injury, poisoning and procedural complications) | 1
Cheilitis (Gastrointestinal disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Chills (General disorders) | 3
Cognitive disturbance (Nervous system disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Confusion (Psychiatric disorders) | 3
Confusion (Gastrointestinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Creatinine increased (Investigations) | 3
Dehydration (Metabolism and nutrition disorders) | 7
Diarrhea (Gastrointestinal disorders) | 17
Dizziness (Nervous system disorders) | 2
Dry mouth (Gastrointestinal disorders) | 2
Dry skin (Gastrointestinal disorders) | 4
Dysgeusia (Nervous system disorders) | 7
Dyspepsia (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Dysuria (Renal and urinary disorders) | 2
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 1
Edema limbs (General disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Fall (Injury, poisoning and procedural complications) | 3
Fatigue (General disorders) | 15
Fecal incontinence (Gastrointestinal disorders) | 1
Fever (General disorders) | 2
Flatulence (Gastrointestinal disorders) | 4
Flushing (Vascular disorders) | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1
Gastroparesis (Gastrointestinal disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Gum infection (Infections and infestations) | 1
Hair color changes (Skin and subcutaneous tissue disorders) | 2
Headache (Nervous system disorders) | 7
Hematoma (Vascular disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Hot flashes (Vascular disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 8
Hypoalbuminemia (Metabolism and nutrition disorders) | 8
Hypocalcemia (Metabolism and nutrition disorders) | 9
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 13
Hypothyroidism (Endocrine disorders) | 3
Infections and infestations - Other (Infections and infestations) | 2
Insomnia (Psychiatric disorders) | 4
Lethargy (Nervous system disorders) | 1
Lung infection (Infections and infestations) | 1
Lymphocyte count decreased (Investigations) | 1
Memory impairment (Nervous system disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 3
Muscle cramp (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 9
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Neutrophil count decreased (Investigations) | 8
Non-cardiac chest pain (General disorders) | 2
Oral pain (Gastrointestinal disorders) | 1
Pain (General disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2
Palpitations (Cardiac disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Paresthesia (Nervous system disorders) | 1
Paronychia (Infections and infestations) | 2
Pelvic pain (Reproductive system and breast disorders) | 1
Platelet count decreased (Investigations) | 16
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3
Psychiatric disorders - Other (Psychiatric disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Rectal pain (Gastrointestinal disorders) | 1
Restlessness (Psychiatric disorders) | 1
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Serum amylase increased (Investigations) | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Syncope (Nervous system disorders) | 1
Thromboembolic event (Vascular disorders) | 2
Thyroid stimulating hormone increased (Investigations) | 4
Tooth infection (Infections and infestations) | 1
Urine discoloration (Renal and urinary disorders) | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Weight loss (Investigations) | 7
White blood cell decreased (Investigations) | 1
Wound infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/10/NCT04197310/Prot_SAP_000.pdf